CLINICAL TRIAL: NCT02014194
Title: Attentional Bias and Attentional Bias Modification Treatment in Obsessive-compulsive Disorder
Brief Title: Attentional Bias Modification Treatment in OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roseli Shavitt (Other)
Responsible Party: Sponsor-Investigator, Roseli Shavitt, MD, Phd, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13674113.2.0000.0068
Record Dates: First submitted 2013-11-25; First posted 2013-12-18 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Obsessive-compulsive Disorder
Keywords: Attentional Bias; Attentional Bias modification treatment
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- attentional bias modification, placebo (Placebo Comparator): Measure of attentional bias modification treatment after 10 sessions of attentional bias modification (two arms). There are two arms with 15 OCD patients each one.
  Interventions: Behavioral: attentional bias modification treatment
- attentional bias modification, active group (Active Comparator): Measure of attentional bias modification treatment after 10 sessions of attentional bias modification (two arms).
  Interventions: Behavioral: attentional bias modification treatment

INTERVENTIONS:
Behavioral: attentional bias modification treatment — The attentional bias modification treatment is a behavioral computerized program (software e-prime)

SUMMARY:
Obsessive-compulsive disorder is a chronic condition. Even with proper treatment, no significant improvement is reached in about 30% to 40% of patients. Thus, the development of new treatment strategies is necessary. The attentional bias - ability to aversive stimuli in capturing the attention of an individual compared to a neutral stimulus - has been extensively studied. Already training attentional bias modification has been shown effective in reducing anxiety present in other anxiety disorders.This project aims to: 1 - generate knowledge on attentional bias in individuals with OCD through the use of a standardized protocol developed for OCD; 2 - available to the scientific community the first specific paradigm for the study of attentional bias in OCD patients, 3 - test the effectiveness of a training protocol for reversing attentional bias in individuals with OCD.

ELIGIBILITY:
Inclusion Criteria: - 30 patients with obsessive-compulsive diagnosis according to DSM-V (with cleaning and or symmetry dimensions)

* 30 health controls

Exclusion Criteria: - doing any kind of behavioral therapy in the moment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of reduction of attentional bias | Patients will be followed an expected average of 7 weeks (baseline, 2 sessions per week - totalizing 5 weeks, 10 sessions and a session after end of treatment). Measures of attentional bias will be assessed in baseline, session 5 and after session 10.

SECONDARY OUTCOMES:
Reduction of anxiety symptoms | Baseline, session 5 and end of treatment (after session 10) (expected average of 7 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo Medical School, São Paulo, Brazil